CLINICAL TRIAL: NCT00979017
Title: Avastin in Combination With Temozolomide and Irinotecan for Unresectable or Multifocal Glioblastoma Multiformes and Gliosarcomas
Brief Title: Avastin/Temozolomide/Irinotecan for Unresectable/Multifocal Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Katy Peters (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Katy Peters, Assistant Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00019065
Record Dates: First submitted 2009-09-15; First posted 2009-09-17 (Estimated); Results first posted 2013-08-12 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-02

CONDITIONS: Glioblastoma Multiforme; Gliosarcoma
Keywords: malignant glioma; glioblastoma multiforme; gliosarcoma; Avastin; bevacizumab; Temodar; temozolomide; Irinotecan; CPT-11; Pro00019065; Vredenburgh; Duke
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma | interventions — Bevacizumab; Temozolomide; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avastin in combination with temozolomide and irinotecan (Experimental): Avastin 10 mg/kg every 14 days. Temozolomide 200 mg/m2 daily x 5 days in a 28-day cycle. Irinotecan dose depends on whether the patient is on an enzyme-inducing antiepileptic drug (EIAED). EIAED 340 mg/m2 every other week and no EIAED 125 mg/m2 every other week. Irinotecan dose also depends on if the patient has the UGT 1A1 polymorphism (7/7). If so, they do not metabolize the irinotecan normally, so these patients will start out at a two dose level reduction. EIAED starting dose will be 275 mg/m2 and no EIAED starting dose will be 75 mg/ m2.
  Interventions: Drug: Avastin; Drug: Temozolomide; Drug: Irinotecan

INTERVENTIONS:
Drug: Avastin — Avastin, by intravenous infusion, 10 mg/kg every 14 days
  Other Names: Avastin (bevacizumab)
Drug: Temozolomide — Oral temozolomide at 200 mg/m2 daily for 5 days
  Other Names: Temodar
Drug: Irinotecan — Irinotecan, by intravenous infusion, every other week (dose dependent upon if taking enzyme-inducing anti-epileptic drugs or if a blood test indicates the patient has the UGT 1A1 polymorphism)
  Other Names: CPT-11, Camptosar

SUMMARY:
The primary objective of the study is to determine the efficacy of Avastin in combination with temozolomide and irinotecan in terms of response rate. The secondary objectives are to describe the overall and progression-free survivals of unresectable patients treated with upfront Avastin, temozolomide and irinotecan and to assess the safety of Avastin, temozolomide and irinotecan in unresectable glioblastoma patients.

This is a phase II study with the combination of Avastin, temozolomide and irinotecan for unresectable or multifocal World Health Organization (WHO) grade IV malignant glioma patients. Patients will receive up to four cycles of Avastin, temozolomide and irinotecan. Approximately 41 subjects will take part in this study at Duke.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of WHO grade IV primary malignant glioma (glioblastoma multiforme or gliosarcoma). Patients will be unresectable or have multifocal disease.
* Age > or = to 18 years and a life expectancy of >12 weeks.
* Evidence of measurable primary Central Nervous System (CNS) neoplasm on contrast enhanced MRI.
* An interval of at least one week between prior biopsy or four weeks from surgical resection and enrollment on this protocol.
* Karnofsky > or = to 60%.
* Hemoglobin > or = to 9g/dl, absolute neutrophil count (ANC) > or = to 1,500 cells/microliter, platelets > or = to 125,000 cells/microliter.
* Serum creatinine ≤ 1.5 mg/dl, serum serum glutamic oxaloacetic transaminase (SGOT) and direct bilirubin ≤ 1.5 times upper limit of normal (if the total bilirubin is greater than or equal to 1.5 x the upper limit of normal, then the direct bilirubin must be ≤ 1.5 x the upper limit of normal).
* Signed informed consent approved by the Institutional Review Board prior to patient entry.
* If sexually active, patients will take contraceptive measures for the duration of the treatments.

Exclusion Criteria:

* Pregnancy or breast feeding
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids.
* Active infection requiring IV antibiotics.
* Treatment with radiotherapy or chemotherapy for a brain tumor, irrespective of the grade of the tumor.
* Evidence of > grade 1 CNS hemorrhage on baseline MRI or CT scan.

Avastin-specific Exclusion Criteria:

* Inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by either urine protein:creatinine (UPC) ratio > or = to 1.0 at screening OR urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of Avastin
* Pregnant (positive pregnancy test) or lactating. Use of effective means of contraception (men and women) in subjects of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-11; Primary Completion 2011-02 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine B Peters, MD, PhD, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Peters KB, Lou E, Desjardins A, Reardon DA, Lipp ES, Miller E, Herndon JE 2nd, McSherry F, Friedman HS, Vredenburgh JJ. Phase II Trial of Upfront Bevacizumab, Irinotecan, and Temozolomide for Unresectable Glioblastoma. Oncologist. 2015 Jul;20(7):727-8. doi: 10.1634/theoncologist.2015-0135. Epub 2015 May 29. PMID 26025933
- See also: The Preston Robert Tisch Brain Tumor Center — http://www.cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Groups:
- Avastin in Combination With Temozolomide and Irinotecan: Avastin 10 mg/kg every 14 days. Temozolomide 200 mg/m2 daily x 5 days in a 28-day cycle. Irinotecan dose depends on whether the patient is on an enzyme-inducing antiepileptic drug (EIAED). EIAED 340 mg/m2 every other week and no EIAED 125 mg/m2 every other week. Irinotecan dose also depends on if the patient has the UGT 1A1 polymorphism (7/7). If so, they do not metabolize the irinotecan normally, so these patients will start out at a two dose level reduction. EIAED starting dose will be 275 mg/m2 and no EIAED starting dose will be 75 mg/ m2.
  Avastin in combination with temozolomide and irinotecan : Avastin, by intravenous infusion, 10 mg/kg every 14 days in combination with oral temozolomide at 200 mg/m2 daily for 5 days and irinotecan, by intravenous infusion, every other week (dose dependent upon if taking enzyme-inducing anti-epileptic drugs or if a blood test indicates the patient has the UGT 1A1 polymorphism)
Period: Overall Study
Arm/Group | Avastin in Combination With Temozolomide and Irinotecan
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Avastin in Combination With Temozolomide and Irinotecan
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: The percentage of participants with a complete or partial response as determined by a modification of the Response Assessment in Neuro-Oncology (RANO) criteria. Complete Response (CR) was defined as complete disappearance on MR/CT of all enhancing tumor and mass effect, off all corticosteroids (or receiving only adrenal replacement doses) and accompanied by a stable or improving neurologic examination. Partial Response (PR) was defined as greater than or equal to 50% reduction in tumor size on MR/CT by bi-dimensional measurement, on a stable or decreasing dose of corticosteroids and accompanied by a stable or improving neurologic examination. Per the criteria, confirmation of response was required. Response rate = CR+PR.
Time Frame: 4 months
Population: Intent-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avastin in Combination With Temozolomide and Irinotecan
Number analyzed (Participants) | 41
percentage of participants | 22 [12 to 37]

2. Secondary Outcome: Incidence and Severity of Central Nervous System (CNS) Hemorrhage and Systemic Hemorrhage
Description: Incidence and severity of CNS hemorrhage and systemic hemorrhage- The adverse events for this study were collected using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, and have been converted to CTCAE version 4.0 for entry into ClinicalTrials.gov.
Time Frame: 4 months
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Avastin in Combination With Temozolomide and Irinotecan
Number analyzed (Participants) | 41
participants
  CNS hemorrhage (grade 3) | 1
  Systemic hemorrhage (all grade 3) | 3

3. Secondary Outcome: Incidence of Grade ≥ 4 Hematologic and ≥ Grade 3 Non-hematologic Toxicities
Description: Incidence of treatment-related, grade ≥ 4 hematologic and ≥ grade 3 non-hematologic toxicities- The adverse events for this study were collected using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, and have been converted to CTCAE version 4.0 for entry into ClinicalTrials.gov.
Time Frame: 4 months
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Avastin in Combination With Temozolomide and Irinotecan
Number analyzed (Participants) | 41
participants
  Grade > or = to 4 hematologic toxicity | 7
  Grade > or = to 3 non-hematologic toxicity | 17

4. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Time in months from the start of study treatment to the date of first progression according to RANO criteria, or to death due to any cause. Per RANO, progression is a ≥ 25% increase in the sum of the products of perpendicular diameters of enhancing lesions, worsening T2/FLAIR, any new lesion, or clinical deterioration. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.
Time Frame: 36 months
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avastin in Combination With Temozolomide and Irinotecan
Number analyzed (Participants) | 41
months | 8.6 [3.5 to 11.3]

5. Secondary Outcome: Median Overall Survival (OS)
Description: Time in months from the start of study treatment to the date of death due to any cause. Patients alive as of the last follow-up had OS censored at the last follow-up date. Median OS was estimated using a Kaplan-Meier curve.
Time Frame: 36 months
Population: Intent-to-treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avastin in Combination With Temozolomide and Irinotecan
Number analyzed (Participants) | 41
months | 12 [7.2 to 13.5]

ADVERSE EVENTS:
Time Frame: 4 months
Description: The adverse events for this study were collected using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, and have been converted to CTCAE version 4.0 for entry into ClinicalTrials.gov.
Arm/Group | Avastin in Combination With Temozolomide and Irinotecan
Serious Adverse Events (participants affected / at risk) | 18/41
Other Adverse Events (participants affected / at risk) | 20/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin in Combination With Temozolomide and Irinotecan (N=41)
Anemia (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 5
Fatigue (General disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Lung infection (Infections and infestations) | 3
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
White blood cell decreased (Investigations) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Intracranial hemorrhage (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 6
Hematuria (Renal and urinary disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin in Combination With Temozolomide and Irinotecan (N=41)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 10
White blood cell decreased (Investigations) | 4
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Confusion (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Thromboembolic event (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes